CLINICAL TRIAL: NCT04063761
Title: Evaluating Active Esophageal Cooling During Cardiac Ablation Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Cooling Therapy, Inc., d/b/a Attune Medical (Industry)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Organization: Advanced Cooling Therapy LLC, d/b/a Attune Medical (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AMEVAB2019
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Results first posted 2022-09-07 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2022-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Esophageal Cooling (Experimental): Single arm study: Patients receive the Attune Medical Esophageal Heat Transfer Device
  Interventions: Device: esophageal cooling device (Attune Medical, Chicago, IL)

INTERVENTIONS:
Device: esophageal cooling device (Attune Medical, Chicago, IL) — Prospective, single center pilot study

SUMMARY:
Left atrial catheter ablation including pulmonary vein isolation is a standard therapy in the management of symptomatic atrial fibrillation; however thermal esophageal injury is a known potential consequence of this procedure. Delivery of radiofrequency (RF) energy necessary to perform left atrial ablation has the potential to cause injury to the nearby esophagus including ulceration, hematoma, spasm, esophageal motility disorders, and, in the most extreme case, atrial-esophageal fistula (AEF). Esophageal mucosal lesions are the likely precursor to AEF, and esophageal mucosal lesions have been detected on post-ablation endoscopy after pulmonary vein isolation with an incidence ranging from 3% to 60%.

Active esophageal cooling during RF ablation as a means of esophageal injury prevention has been investigated through mathematical models, pre-clinical studies, and in clinical trials. Existing data support the efficacy of this approach, but the practice has not been widely adopted due to lack of a commercially available device.

The aim or purpose of this study is to evaluate the impact on procedural efficiency of ablation procedures performed using esophageal heat transfer to cool the esophagus during left atrial RF ablation.

DETAILED DESCRIPTION:
This study is a prospective, pilot study using the Attune Medical esophageal heat transfer device to actively cool the esophagus during RF ablation procedures. This design is appropriate to gather the data needed regarding overall procedural time, compare this to historical controls, and estimate a sample size for a larger study powered for statistical significance.

The subjects will undergo preparation and anesthesia procedures following standard practice. Once the patient is intubated, the esophageal heat transfer device will be placed into the esophagus according to the Instructions for Use (IFU). The device will remain in place until the ablation procedure is completed and will be removed before extubation. Posterior left atrial wall ablation using standard parameters will only be performed when the esophageal heat transfer device has reached a temperature of 4-6 degrees C for at least 2 minutes. The device will be set to neutral or warming temperature (37-42 degrees C) during other aspects of the procedure (such as mapping and anterior wall ablations).

All patients will be followed up in total for 6 weeks (Long Term Follow-up visit) after the procedure to document any clinical complication related to thermal esophageal injuries if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age over 18 years)
* Undergoing first left atrial ablation for the treatment of atrial fibrillation (AF) including pulmonary vein isolation
* Undergoing catheter-based ablation procedure using radiofrequency energy
* Patients must be able to understand and critically review the informed consent form.
* Subjects must understand and agree to study requirements and sign a written informed consent.

Exclusion Criteria:

* Patients who are unable to provide informed consent.
* History of prior atrial fibrillation (AF) ablation procedures.
* Significant co-morbidities that preclude standard ablation procedure.
* Patients with <40 kg of body mass
* Patients with relevant esophageal pathology (e.g. esophageal cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Mazur, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Esophageal Cooling
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Esophageal Cooling
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Total Time of Active Ablation Procedure
Description: Study Day 1 for all patients enrolled, during left atrial ablation procedures using radiofrequency energy, up to 5 hours. Measured as total procedure time as documented by clinician recorder and research coordinator.
Time Frame: Study Day 1 for all patients enrolled, during left atrial ablation procedures using radiofrequency energy, up to 5 hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Esophageal Cooling
Number analyzed (Participants) | 20
Hours | 3.26 (0.7)

2. Secondary Outcome: Total Procedure Time
Description: Study Day 1 for all patients enrolled, during left atrial ablation procedures using radiofrequency energy, up to 5 hours after procedure. Measured as total procedure time to discharge to PACU as documented by clinician recorder and research coordinator.
Time Frame: Study Day 1 for all patients enrolled from patient entry to Electrophysiology (EP) lab until post procedure discharge to Post-Anesthesia Care Unit (PACU)
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Esophageal Cooling
Number analyzed (Participants) | 20
Hours | 5.11 (0.59)

3. Secondary Outcome: Number of Procedural Pauses During Left Atrial Instrumentation
Description: Number of procedural pauses during left atrial instrumentation measured from trans-septal puncture to achievement of Pulmonary Vein Isolation (PVI)
Time Frame: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Procedural pauses
Arm/Group | Esophageal Cooling
Number analyzed (Participants) | 20
Procedural pauses | 0 [0 to .168]

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Esophageal Cooling
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT04063761/Prot_SAP_000.pdf